CLINICAL TRIAL: NCT00698178
Title: Waist Circumference Versus Body Mass Index to Predict Severity of Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Hsin-Hong Chen/Superintendent, Lotung Poh-Ai Hospital
Other Study IDs: OMCP-97-009
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Gastroesophageal Reflux Disease; Obesity
Keywords: Gastroesophageal reflux disease; Waist circumference; Body mass index; Obesity
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- NERD: patients with typical gastro-reflux symptoms but no erosions were discernible on upper gastrointestinal endoscopy
  Interventions: Other: Anthropometric measurements
- EE: Patients with both typical gastroesophageal reflux symptoms and characteristic flam-like erosions as demonstrated on upper gastrointestinal endoscopy
  Interventions: Other: Anthropometric measurements
- FD: Patients report no typical reflux symptoms but fulfill diagnostic criteria of functional dyspepsia, whose upper gastrointestinal endoscopy are negative.
  Interventions: Other: Anthropometric measurements

INTERVENTIONS:
Other: Anthropometric measurements — All patients undergo anthropometric measurements to record body weight, body height and waist circumference on the day of enrollment

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common and important disorder. Previous studies have demonstrated the association of obesity with GERD, and now obesity is regarded as a risk factor for GERD. Moreover, body mass index (BMI), an indicator of general obesity, correlates with severity of symptoms and degree of erosive esophagitis. Waist circumference, an indicator of abdominal obesity, has stronger correlation with intra-abdominal pressure and low-grade inflammatory state when compared with BMI. Nevertheless the association of waist circumference with severity of GERD has not been studied.

The primary aim of this study is to compare BMI with waist circumference for their independent association with severity of GERD. The secondary aim is to evaluate independent risk factors of severity of GERD.

DETAILED DESCRIPTION:
This is a cross-section observational study. Outpatients presenting with acid reflux or heart burn are interviewed with standardized questionnaire to quantify severity of symptoms. The eligible patients undergo upper endoscopy to diagnose erosive esophagitis and further classify the degree of erosions according to Los-Angels classification. Enrolled patients receive anthropometric measurements to record body weight, body height and waist circumference on the day of enrollment.

Two outcomes are studied: the severity of GERD symptoms and the Los-Angels Classification of erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years old and less than 70 years old
* typical gastroesophageal reflux symptoms (heart burn and acid reflux)
* outpatient
* complete upper gastrointestinal endoscopy

Exclusion Criteria:

* age less than 20 years or more than 70 years old
* receive medication for reflux disease (including proton pump inhibitor, histamine type 2 receptor blocker, prokinetic agents) in previous one month
* pregnant women
* history of abdominal surgery
* severe comorbidity with cirrhosis, end-stage renal disease, heart failure
* no written informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients at a general hospital with 1000 beds in north-eastern Taiwan
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
the degree fo erosive esophagitis according to Los-Angels classification | on the day of endoscopy examination

SECONDARY OUTCOMES:
gastro-reflux severity score as evaluated by standardized questionnaire | at enrollment (before upper GI endoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chun Hsu, M.D., Principal Investigator — Lotung Poh-Ai Hospital, Ilan, Taiwan
Locations (1):
- Lotung Poh-Ai Hospital, Lotung Town, Ilan County, Taiwan